CLINICAL TRIAL: NCT02916563
Title: Dario Blood Glucose Monitoring System - Android Devices Altitude Evaluation
Brief Title: Dario Blood Glucose Monitoring System - Android Devices Altitude Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-0006
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude (Experimental): Single arm study Blood Glucose Monitoring System Altitude Performance
  Interventions: Device: Blood Glucose Monitoring System Altitude Performance

INTERVENTIONS:
Device: Blood Glucose Monitoring System Altitude Performance — Performance as assessed against a reference method at an altitude of approximately 10,000 feet.

SUMMARY:
This study evaluates the performance of a blood glucose monitoring system at high altitudes (approximately 10,000 feet). The performance is assessed via a reference method for glucose analysis (Yellow Springs Instrument 2300 STAT Plus Glucose Analyzer).

DETAILED DESCRIPTION:
This study will be a non-randomized study conducted to assess the accuracy and performance of the Dario Blood Glucose Monitoring System at an elevated altitude. 50 subjects will be enrolled in this study. Participation includes a 15-20 minute visit to the clinical site where they will be consented. The participant will then receive a fingerstick to obtain capillary blood used to test the performance of the BGMS and to obtain a comparative glucose measurement on the reference method, the Yellow Springs Instrument 2300 STAT Plus Glucose Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English

Exclusion Criteria:

* Pregnant
* Has any condition that the principle investigator believes may interfere in the subject's participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Individuals With Type 1 or Type 2 Diabetes and Individuals Without Diabetes: A total of 50 subjects diagnosed with type 1 or type 2 diabetes and individuals without diabetes.
  1. Age of subject is 18 years or older
  2. Able to speak and read English
Period: Overall Study
Arm/Group | Individuals With Type 1 or Type 2 Diabetes and Individuals Without Diabetes
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Individuals With Type 1 or Type 2 Diabetes and Individuals Without Diabetes
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Glucose Readings
Description: The success criterion for the performance of the Blood Glucose Monitoring System at high altitude (approximately 10,000 feet above sea level) means that 95% of the blood glucose readings fall within 15mg/dL of the YSI reference value (for reference values less than 75 mg/dL) and within 20% (for reference values greater than or equal to 75 mg/dL).
Time Frame: One day
Population: Each subject will be measured 9 times with the Dario system: 3 strips lots for each of the three representative smart mobile devices (total of nine meters) under evaluation (150 strips per mobile device, total no. of strips 450).
Measure: Number; unit: Number of Glucose readings in range
Units Other Than Participants: Glucose readings
Arm/Group | Individuals With Type 1 or Type 2 Diabetes and Individuals Without Diabetes
Number analyzed (Participants) | 50
Number analyzed (Glucose readings) | 450
Number of Glucose readings in range | 449

ADVERSE EVENTS:
Time Frame: The study was performed during one day
Arm/Group | Altitude
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes